CLINICAL TRIAL: NCT02139553
Title: Effect of Rhythmic Upper-limb Training in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ULRM-001
Record Dates: First submitted 2014-04-30; First posted 2014-05-15 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Cerebral Stroke
Keywords: Rhythmic versus discrete movements; Rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rhythmic rehabilitation (Experimental): Patients undergo a first evaluation, and a second evaluation one month later to determine their natural evolution. The following month, patients get 12 sessions of rhythmic therapy. A third evaluation is organized straight after this month and a fourth evaluation, 3 months after to assess the after-effects of the therapy.
  Interventions: Procedure: Rhythmic rehabilitation

INTERVENTIONS:
Procedure: Rhythmic rehabilitation — Stroke patients have 12 rehabilitation sessions on a planar rehabilitation robot, Reaplan, focussed on rhythmic arm movements.

SUMMARY:
The purpose of this study is to determine whether rhythmic upper-limb movement training in post-stroke patients allows to improve only this particular type of movements or if it also improves some parameters of discrete movements. Based on our results we hope to be able to answer a fundamental question: are rhythmic and discrete movements two independent primitives?

DETAILED DESCRIPTION:
Patients are assessed four times during this longitudinal study. One month separates the first two assessment, next patients are trained 12 times during one month with rhythmic movement training on an end-effector robot. After this month, patients are assessed a third time and three months later a fourth time in order to study long-time benefits of the therapy.

ELIGIBILITY:
Inclusion Criteria:

* more than 6 months post-stroke patients
* Fugl-Meyer between 7 and 55
* Maintain the same intensity of rehabilitation during the study

Exclusion Criteria:

* cerebellar stroke
* severe aphasia or cognitive disorder
* any other neurological disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2014-10 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in movement smoothness in rhythmic straight movements after one month of rhythmic therapy | 1 week to 1 day before therapy and 1 day to 1 week after therapy
  Patients are asked to fulfill rhythmic movements on the end-effector robot Reaplan. The smoothness is assessed with following metrics:
  * number of peaks in velocity profile
  * TENT value
  * logarithmic dimensionless square jerk
Change in movement smoothness in discrete straight movements after one month of rhythmic therapy | 1 week to 1 day before therapy and 1 day to 1 week after therapy
  Patients are asked to fulfill discrete movements on the end-effector robot Reaplan. The smoothness is assessed with following metrics:
  * number of peaks in velocity profile
  * TENT value
  * logarithmic dimensionless square jerk
Change in accuracy of discrete straight movements after one month of rhythmic therapy | 1 week to 1 day before therapy and 1 day to 1 week after therapy
  Patients are asked to fulfill discrete movements on the end-effector robot Reaplan. The accuracy is assessed.
Change in smoothness of rhythmic circular movement after rhythmic therapy | 1 day to 1 week before therapy and 1day to 1 week after therapy
  Patients are asked to fulfill 10 circular movements on the end-effector robot Reaplan. The movement smoothness are assessed

SECONDARY OUTCOMES:
Change of the general motricity of the patient due to one month rhythmic therapy | 1 week to 1 day before therapy and 1 day to 1 week after therapy
  1. Upper limb Fugl-Meyer Assessment
  2. Box and block test
  3. Ashworth test
Therapy after effects | 1 day to one week after therapy and 3 months after therapy
  Evolution of the movement smoothness in rhythmic and discrete movements, the movement accuracy in discrete movements and the general motricity
Assessment of the natural evolution of the patient | 4 to 5 weeks before therapy and 1 week to 1 day before therapy
  Natural evolution of the movement smoothness in rhythmic and discrete movements, of the accuracy in discrete movements and of the general motricity of the patient

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques universitaires Saint-Luc, Woluwe-St-Lambert, Brabant Wallon, Belgium

IPD SHARING:
Plan to Share IPD: Undecided